CLINICAL TRIAL: NCT05606471
Title: The Anabolic Effects of GLP-1 Agonism to Prevent Lean Muscle Losses During Very-low Calorie Diets (VLCDs) for Weight Loss
Brief Title: Glucagon-like Peptide-1 Agonism With Very Low Calorie Diets
Acronym: SemVLCD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21031
Record Dates: First submitted 2022-05-23; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes Mellitus in Obese
Keywords: Type 2 diabetes; Obesity; GLP-1; Semaglutide; VLCD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VLCD only (Active Comparator): Participants in this group will be placed on a very-low calorie diet with a daily energy intake limit of 800 kilocalories. 600 kilocalories will be made up of total meal replacement products supplied by Lighterlife UK. The remaining 200 kilocalories will be flexible for participants to add additional vegetables to supplement the total meal replacement products, allowing some variety to the diet.
  Interventions: Dietary Supplement: Very-low Calorie Diet
- Semaglutide only (Active Comparator): Participants will be asked to self-administer the GLP-1 agonist Semaglutide weekly, as per clinical practice. They will be asked to start at 0.25mg and increase every two weeks (if tolerated) to the maintenance dose of 1mg, which they will continue until the end of the study.
  Interventions: Drug: Semaglutide Pen Injector [Ozempic]
- Combined VLCD plus Semaglutide (Experimental): Participants in this group will both partake in the VLCD, and take the weekly dose of Semaglutide (as described above).
  Interventions: Drug: Semaglutide Pen Injector [Ozempic]; Dietary Supplement: Very-low Calorie Diet

INTERVENTIONS:
Drug: Semaglutide Pen Injector [Ozempic] — Glucagon-like peptide 1 (GLP-1) receptor agonist
  Arms: Combined VLCD plus Semaglutide; Semaglutide only
Dietary Supplement: Very-low Calorie Diet — Total meal replacement with a limit of 800 kilocalories per day
  Arms: Combined VLCD plus Semaglutide; VLCD only

SUMMARY:
The very-low calorie diet (VLCD) is a highly effective and safe way to rapidly lose significant amounts of weight and dramatically improve blood sugar control in a short period of time (typically 8-12 weeks). It has recently become recommended by the UK National Health Service as a treatment for selected patients with type 2 diabetes. One drawback of VLCD however is the associated loss of skeletal muscle which affects some patients.

Semaglutide is a well-known medication for type 2 diabetes that also improves blood sugar control and facilitates weight loss. Recent research has shown that it may also stimulate muscle growth, meaning it could help to preserve muscle mass during weight loss. Therefore, this research study aims to see whether taking Semaglutide alongside the VLCD reduces the amount of muscle lost, and could improve the long-term outcomes of VLCD.

The study will take place in the Medical School building in the Royal Derby Hospital. Up to 45 participants will be recruited and allocated into one of 3 groups:

1. Semaglutide only
2. VLCD only
3. Combined Semaglutide plus VLCD The study is 12 weeks in duration and consists of four visits including two 6-hour visits, one 4-hour visit and one 30-minute visit. The first visit is a short Preliminary Visit where participants are asked to ingest stable isotope drinks for measurement of muscle growth rates and muscle mass. Food intake and physical activity monitoring will also be commenced.

Visits 1 & 3 are identical and occur at the beginning and end of the 12-week intervention period, respectively. During these visits participants will undergo a Dual-energy X-ray absorptiometry (DXA) scan, a right vastus lateralis muscle ultrasound scan & muscle biopsy, an intravenous glucose tolerance test, electromyography, tests of muscular function, gait & balance, and questionnaires regarding quality of life & physical activity. These visits are expected to last up to 6 hours.

Visit 2 is a shorter visit mid-way through the 12 weeks, lasting approximately 4.5 hours. Participants will undergo another DXA scan and muscle biopsy in addition to having multiple blood tests taken over a 4-hour period to determine muscle protein breakdown rates.

During the 12 weeks, those in the VLCD group will be asked to stick strictly to an 800 kilocalorie very-low calorie diet, whilst those in the Semaglutide group will be required to inject themselves with Semaglutide once a week. Those in the combined group will be asked to do both. All participants will be monitored closely throughout the 12-week period, with regular phone calls and/or emails.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Type 2 Diabetes Mellitus
* Body mass index > 27kg·m-2
* Eligible for VLCD, Semaglutide (or both), within routine practice
* Ability to provide informed consent

Exclusion Criteria:

* BMI > 50kg·m-2
* Current pregnancy or breastfeeding, or intention to fall pregnant within the next 3 months
* Uncontrolled hypertension (blood pressure >200/120mmHg)
* Current treatment with insulin
* Current or recent use of GLP-1 agonists
* Previous adverse reaction to a GLP-1 agonist
* Current or recent involvement in a VLCD programme (within the last 12 months)
* History of >5% weight loss within the preceding 12 months
* Ingestion of exogenous D2O within the preceding 12 months
* Background of clinically significant cardiovascular, cerebrovascular or respiratory disease, neurological disorders or musculoskeletal problems
* History of malignancy undergoing current treatment or palliation
* History of any medical condition contraindicating the use of GLP-1 agonist medication
* Any other medical condition deemed by the investigators to preclude inclusion into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-07-28 (Estimated); Study Completion 2023-07-28 (Estimated)

PRIMARY OUTCOMES:
Muscle protein synthesis rate | 6 weeks
  Measuring the rate of skeletal muscle growth in vivo by determining the rate of deuterium incorporation into muscle
Muscle protein breakdown rate | 6 weeks
  Measuring the rate of breakdown of skeletal muscle in vivo using the rate of appearance of deuterium-labelled 3-methyl-histidine in blood after an initial oral bolus

SECONDARY OUTCOMES:
Skeletal muscle mass | 12 weeks
  Determined from DXA scanning (measured in kg and percentage of total body weight) and novel techniques using rate of appearance of a creatine tracer in urine after an initial bolus
Fat mass | 12 weeks
  Determined from DXA scanning (measured in kg and percentage of total body weight)
Total body weight | 12 weeks
  Measured in kg
Whole body insulin sensitivity | 12 weeks
  Determined using the intravenous glucose tolerance test and measures of fasting insulin & glucose
Pancreatic beta cell function | 12 weeks
  Determined using the intravenous glucose tolerance test and measures of fasting insulin & glucose
Skeletal muscle strength | 12 weeks
  Determined from maximal voluntary contraction (MVC) of left knee extension
Skeletal neuromuscular function | 12 weeks
  Assessed using measurement of force stability during electromyography
Gross skeletal muscle function | 12 weeks
  Measured using a short battery of physical performance tests (SBPPT) to give an overall score of skeletal gross skeletal muscle function (scored out of 12)
Right vastus lateralis muscle thickness | 12 weeks
  Determined from muscle ultrasonography
Right vastus lateralis muscle cross sectional area (CSA) | 12 weeks
  Determined from muscle ultrasonography
Right vastus lateralis muscle fibre pennation angle | 12 weeks
  Determined from muscle ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Iskandar Idris, Principal Investigator — Professor in Diabetes and Vascular Medicine & Honorary Consultant
Locations (1):
- University of Nottingham, Royal Derby Hospital Centre, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No